## **VA INFORMED CONSENT PROCESS CHECKLIST**

\*Complete this checklist for each consent obtained and file with the original informed consent document\*

| RESEARCH STUDY IDENTIFICATION (Required information) |
|---|
| STUDY TITLE: Link Up: Facilitating use of the Veterans Crisis Line in High-Risk Patients |
| PI:Mark Ilgen, PhD |
| NAME OF STUDY TEAM MEMBER OBTAINING CONSENT: |
| ROLE OF STUDY TEAM MEMBER OBTAINING CONSENT: |

ORIGINAL FORM VERSION: 4/15/09. REVISIONS: 9/17/09, 10/30/09, 11/30/09, 12/07/11, 2/27/12, 10/7/13

| RESI | EARCH SUBJECT IDENTIFICAT | ION: (Requir | ed information) | | |
|---|---|---|---|---|---|
| | | | 1 1 1 | 1 1 | |
| Last Name | First Name | Mid. Init. | Last-4 SSN | Todays Date (mm/dd/yy) | _ |

| _ | |
|---|---|
| A. | Date ALL required SIGNATURES (Subject, Witness (If required by IRB) and Person Obtaining Consent), their PRINTED NAMES and the DATES they signed the informed consent document |
| | (ICD) have been Checked and Verified Accurate and appear in the proper location |
| В. | DATE AND TIME (ICD) WAS REVIEWED AND DEEMED COMPLETE AND VALID **Must be prior to date/time of Subject's First Study Activity** |
| C. | DATE AND TIME OF THE SUBJECT'S FIRST STUDY ACTIVITY OR INVOLVEMENT |
| | Verify and Initial each requirement below. |
| 1. | Informed consent and HIPAA Authorization, if required by VA-IRB was obtained from this subject prior to study participation. |
| 2. | A VA Scope of Practice Form has been signed by the PI and approved by the VA IRB which designates me as an authorized agent of the PI and qualified to obtain consent for this study. |
| 3. | This prospective subject was given adequate time necessary to carefully and fully read the Informed consent document (ICD) and all questions were answered to his/her satisfaction. |
| 4. | All aspects of this subject's study involvement, including the purpose of the study, known and potential risks, possible benefits and alternatives to study participation were explained and discussed prior to subject signing the ICD. |
| 5. | If required, a scanned image of the Research Enrollment Note, Consent Form and/or HIPAA Authorization will be entered into the subject's electronic medical record (CPRS). |
| 6. | Subject has been consented using the most recently approved, VA date-stamped version of the consent form (VA Form 10-1086) and HIPAA Authorization Form (VA Form 10-0493). |
| 7. | A copy of the completed and signed, original informed consent document has been issued to this subject and the subject was instructed to retain that copy for reference and to ask any and all questions that might arise throughout their study involvement. |
| 8. | The subject has been shown where in the ICD to locate study team phone number(s) and the phone number of the VAAAHS IRB Coordinator. The subject has been reminded to call with any questions or concerns. Cathy Kaczmarek @ 734.845.3439 |
| 9. | The subject has been informed that participation is entirely voluntary and that they may withdraw their participation at any time and for any reason. |
| 10. | Original ICDs and all copies are printed and issued as single-sided documents and that the original signed ICD must be kept in the investigator's project files on VA property. |
| 11. | Upon completion of the Informed Consent Process, this subject's name was added to the Master List of All Subjects. [Per revised VHA Handbook 1200.05 (11/12/14) a MLS is no longer required, but a list of all enrolled participants is considered good research practice.] |
| 12. | I know I can contact the VAAAHS IRB Coordinator at 734.845.3439 or the Research Compliance Officer at 734.845.3766 if I have questions or concerns regarding the consent of this or any individual considering study participation. |



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: Mark Ilgen, PhD

VAMC: VA Ann Arbor

Healthcare System

**Version Date:** 06/09/2016

## **PURPOSE OF RESEARCH STUDY:**

The purpose of the study is to learn about Veterans who use the Veterans Crisis Line during a suicidal crisis and those who don't. We would also like to learn whether or not Veterans who have experienced a suicidal crisis could benefit from participating in a discussion about their thoughts and perceptions of the Veterans Crisis Line. You have been invited to participate in this research study because you are a patient in this VA psychiatry inpatient unit and were identified as having experienced a suicidal crisis (i.e. recent suicide attempt, significant suicidal thoughts). This is a joint study between the Battle Creek and Ann Arbor VA facilities.

### **DESCRIPTION:**

This is a two part study. Part 1 involves completing a survey only. Based on some of your answers you may be eligible to participate in Part 2. Below is more detail about Part 1 and Part 2:

Part 1: We plan to enroll up to approximately 1042 patients for Part 1 – Screening of this study. If you decide to participate, we will ask you to complete a screening survey, which will take approximately 15-30 minutes. The survey asks questions about topics such as your thoughts and behaviors related to suicide, overall mental health and physical functioning, and your utilization of treatment services, such as the Veterans Crisis Line. Depending on your answers to the screening survey, you may be eligible to participate in the full study (Part 2). If you are found not eligible for participation in the full study, then your participation will be complete at the end of Part 1 and you will have no further contact with our research staff.

Part 2: We plan to enroll approximately 500 patients for Part 2 of this study. If you are eligible and decide to participate in the full study, you will be asked to complete the following:

Baseline Assessment: The baseline assessment will take approximately 45-60 minutes to complete. We will ask questions about topics such as suicide, drug and alcohol use, treatment and service utilization, and perception of those services. You will complete part of the assessment yourself by answering questions on a paper survey and the other part will include interview questions asked by research staff.

*Intervention session:* After completing the baseline assessment you will be randomly placed into one of two groups (assigned by chance in a process similar to "flipping a coin"):

<u>Group 1</u>: If you are in Group 1, you will be asked to participate in a 30-45 minute one-on-one intervention session with a member of our study team to discuss the Veterans Crisis hotline. These sessions will be audio recorded and reviewed by research staff for training purposes and to ensure that the research team is following protocol (making sure that all research team members conduct the sessions in the same way).

<u>Group 2</u>: If you are in Group 2, you will be asked to participate in a brief discussion with a member of our study team, and you will receive informational materials about the Veterans Crisis Line.

Afterwards both groups will be asked to answer some additional questions, which will take approximately 5-10 minutes.

| RESEARCH SUBJECT IDENTIFIC | CATION: (Required infor | mation) | | |
|---|---|---|---|---|
| | | | 1 1 1 | 1 1 |
| Last Name | First Name | Mid. Init. | Last-4 SSN | Todays Date (mm/dd/yy) |
| VA Form 10-1086 | Page 1 | of 5 | | |



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: Mark Ilgen, PhD

VAMC: VA Ann Arbor

Healthcare System


Follow-Up Assessments: Study staff still will contact you to schedule your follow up assessments at about 3, 6, and 12-months after study enrollment. These follow-up sessions will usually take approximately 45-60 minutes. The assessments will ask similar questions as the baseline assessment

Your total participation in Part 2 of the study (i.e. baseline survey, intervention, and 3 follow-up surveys) is expected to occur over a period of approximately 12 months. After you complete the study, we may contact you for an additional interview to ask about your study experience. If you choose to participate in the interview, you will sign a separate consent form for that part.

#### RISKS:

You may experience some discomfort when answering questions, such as questions regarding your experiences with suicide and suicidal thoughts. This type of discomfort is expected to be temporary. You may choose not to answer any questions that make you uncomfortable or that you do not wish to answer.

Another risk is potential loss of confidentiality of some of your personal information. We may be required to break confidentiality if we believe that there is a risk of harm to yourself or someone else (for example, you may harm yourself, someone else, or someone is harming you, or in cases of child or elder abuse). This means that we may be required to inform your regular care providers or authorities to protect you or others. The information we disclose will be relevant to your care and may have been information we obtained during the research, such as your thoughts to harm yourself, your name, and contact information,

As with any research study, there may be other risks that are unforeseeable at this time.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under the following circumstances: if you disclose intent to hurt yourself, others, or if you are being hurt.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to get research information, then the researchers may not use the Certificate to withhold that information.



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: Mark Ilgen, PhD VAMC: VA Ann Arbor

Healthcare System


Being in more than one research study at the same time, or even at different times, may increase the risks to you. It may also affect the results of the studies. You should not take part in more than one study without approval from the researchers involved in each study.

### **BENEFITS:**

Your participation may help us discover how to improve services for veterans in the future. If you participate in Part 2, you may find that participating in this study helps you to learn about options you may have for obtaining help when in a suicidal crisis. However, we cannot and do not guarantee or promise that you will benefit by participating in this study.

## **ALTERNATE COURSES OF ACTION:**

You do not have to participate in this study. You may withdraw from the study at any time without penalty. By doing so, you will not lose any benefits that you may be entitled to. If you choose not to participate in this study, your decision will not affect your eligibility to receive standard health care at the Ann Arbor VAMC.

#### STATEMENT OF RESEARCH RESULTS:

Research data collected as part of this study will be stored according to the privacy and security guidelines established by the VHA. Only authorized research staff will have access to your research data and research files. These authorized research staff may have access to viewing your paper forms and medical records. If you participate in Part 2, authorized research staff may also access your medical records to obtain your contact information to schedule and conduct follow-up appointments. Your name and other identifying information (consent form) will be stored separately from research data (e.g. survey and interview answers). Unique ID numbers will be substituted for names to protect your identity in the data file. Data on paper will be stored in locked filing cabinets at Ann Arbor VA research offices. All electronic study data will be kept in restricted access files and stored on the VA network server. Paper files may be stored on the secure network drive as a PDF. Because this is a joint study between the Battle Creek VAMC and Ann Arbor VAMC, electronic data may be shared/transmitted through the use of VAMC secure servers at either site.

If you participate in Part 2, the audiotapes of the sessions will be converted into computer files and stored on secure servers. Audio-records will be used to evaluate the research staff who are leading the sessions. Audio computer files will be confidential and access will be limited to authorized research staff.

Researchers from the Battle Creek Health Care System and the Ann Arbor VA Health Care System will analyze the data collected from this study. If the results of this study are reported in medical journals or at meetings, you will not be identified by name, by recognizable photograph, or by any other means without your specific consent. No information by which you can be identified will be released or published unless required by law. We will let you know of any important discoveries made during this study which may affect you, your condition, or your willingness to participate in this study.

#### SPECIAL CIRCUMSTANCES:

There will not be any costs to you for any additional care that you receive as a participant in this research study. The investigators of this study may have to end your participation in this study for reasons such as if it is in your best interest; you do not follow the study plan (e.g., do not complete the survey); the investigator decides that continuation could be harmful to you; the study is canceled; other administrative reasons; or other



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: Mark Ilgen, PhD VAMC: VA Ann Arbor

Healthcare System


unanticipated circumstances. If you are withdrawn from the study, it will not affect the treatment you receive from your providers at the Ann Arbor VAMC.

### **COMPENSATION:**

For participating in Part 1, you will receive a \$10 gift card after completing the screening survey.

If you are eligible after screening, and you choose to participate in Part 2, you will receive a \$25 gift card for completion of the baseline assessment and a \$30 gift card for each 3, 6, and 12 month follow-up assessment completed. Therefore, your maximum compensation for this part of the study could be \$115.



| Title of Study: | Link Up | Facilitating Use of the Veterans Crisis Line | | |
|---|---|---|---|---|
| Principal Investig | gator: | Mark Ilgen, PhD | VAMC: | VA Ann Arbor<br>Healthcare System |
| Version Date: | Version Date: 06/09/2016 | | | |
| RESEARCH SUB | JECT'S | | | |
| treatment have bee | has explained this research study and answered all questions. The risks or discomforts and possible benefits of the study have been described. Other choices of available reatment have been explained. Some veterans are required to pay co-payments for medical care and services provided by VA. These co-payment requirements will continue to apply for VA care and services that are not part of this study. | | | |
| no penalty or loss o<br>time without penalty<br>accordance with ap<br>injured by participat<br>been made for addi-<br>medical care and se<br>care and services p | f rights to<br>or loss of<br>plicable for<br>ion in this<br>tional cor<br>ervices provided b | entirely voluntary. You may refuse to particip<br>which individuals are entitled. Participants<br>of VA or other benefits. VA will provide treat<br>ederal regulations. The VA will provide necessisted. You will be treated for the injury at a<br>enpensation. You may be among the veterant<br>covided by VA. These co-payment requirements by VA that are not part of this study. You have<br>gents from liability for negligence by signing | may withdr<br>ment for re-<br>essary med<br>no cost to y<br>s required t<br>ents will cor<br>e not waive | aw from this study at any search related injury in ical treatment should you be ou, but no provisions have to pay co-payments for attinue to apply to medical |
| research study, you<br>3646 during the day<br>on call can be conta | can cont<br>and or pacted at 7<br>255), and | oblems, an injury, or if you have questions, of<br>tact member(s) of the research study team:<br>paged after hours at 734-936-6266 (then dial<br>34-769-7100 after hours. At any time, you not<br>press "1" to connect to a free, 24-hour VA has<br>stration. | Mark Ilgen<br>page ID: 1<br>nay call the | can be called at 734-845-<br>5912) or the VA psychiatrist<br>Veterans Crisis Hotline at |
| research subject an study staff are not a | d to verify<br>vailable o | nan Studies coordinator at 734-845-3440 to<br>y this study is reviewed and approved by the<br>or to discuss your questions or concerns with<br>rch at the VA Ann Arbor Healthcare System | e VA. You n<br>n someone | nay also call when research other than study staff. You |
| I have been informe<br>I will receive a signe | ed about red copy o | my rights as a research subject, and I volunt f this consent form. | arily conse | nt to participate in this study. |
| xSignature of Subject | t | X<br>(Print Name) | | X<br>Todays Date (mm/dd/yy) |
| XSignature of person<br>(Study personnel must b | e approve | | | X Todays Date (mm/dd/yy) IVELY NUMBERED. |
| VA Form 10-1086 [VALID ONLY WITH CURF | | Page 5 of 5 | | |

| Department of Veterans Affairs Authorization for Use and Information Collected for | d Release of Individually Ide<br>VHA Research | ntifiable Health |
|---|---|---|
| Subject Name (Last, First, Middle Initial): | Subject SSN (last 4 only): | Date of Birth: |
| VA Facility (Name and Address): VA Ann Arbor Healthcare System 2215 Fuller Rd. Ann Arbor, MI 48105 | | |
| VA Principal Investigator (PI): | PI Contact Information: | |
| Mark Ilgen, Ph.D. | Mark.Ilgen@va.gov; 734-845-3646 | Ó |
| Study Title: | | |
| Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients | | |
| The purpose of the study is to learn about Veterans who use the Veterans Crisis Li also like to learn whether or not Veterans who have experienced a suicidal crisis or member of our study team about their thoughts and perceptions of the Veterans Cr research study because you are a patient in this VA psychiatry inpatient unit and w recent suicide attempt, significant suicidal thoughts). Based on your responses provinvited to participate in further research activities, including further surveys, interv (Part 2). This is a joint study between the Battle Creek and Ann Arbor VA facilities. | bould benefit from participating in a disis Line. You have been invited to prere identified as having experienced wided during the screening survey (Priews and a discussion with a member | barticipate in this a suicidal crisis (i.e. art 1), you may be |
| USE OF YOUR INDIVIDUALLY IDENTIFIABLE HEALTH INFORM | MATION (IIHI): | |
| Your individually identifiable health information is information about information that would identify you such as your name, date of birth to allow the VA Principal Investigator (PI) and/or the VA research to present health information in addition to new health information the investigators of this study are committed to protecting your privacy your health care. | າ, or other individual identifiers<br>eam members to access and ເ<br>v mav collect for the study nar | . VHA is asking you<br>ise your past or<br>ned above. The |
| Signing this authorization is completely voluntary. However, your are participate in this study. Your treatment, payment, enrollment, or elewhether or not you sign this authorization. | igibility for VA benefits will not | be affected, |
| Your individually identifiable health information used for this VA stu | dy includes the information ma | arked below: |
| | progress notes, medications, | lab or radiology |
| Specific information concerning: | | |
| $oxed{oxed}$ alcohol abuse $oxed{oxed}$ drug abuse $oxed{oxed}$ sickle cell | anemia 🔲 HIV | |
| □ Demographic Information such as name, age, race | | |
| ☐ Billing or Financial Records | | |
| <ul> <li>☑ Questionnaire, Survey, and/or Subject Diary</li> <li>☑ Other as described: We will only access information concerning alcohol or</li> </ul> | or drug abuse for participants in Part | 2. |

**Version Date:** 06/09/2016 Page 1

| Veterans Health Administration (VHA) Research Subject Name (Last, First, Middle Initial): Subject SSN (last 4 only): Date of Birth: |
|---|
| Subject Name (Last, First, Middle Hillar). Subject Son (last 4 Only). Date of Birth. |
| USE OF YOUR DATA OR SPECIMENS FOR OTHER RESEARCH: (Instruction: When banking or further analysis is an optional research activity, complete page 5 and leave this section blank. If banking is a required research activity to store "Data" and/or "Specimen" for future use or if "Not Applicable" is selected, remove page 5 in its entirety.) |
| An important part of this research is to save your |
| □ Data |
| ☐ Specimen |
| in a secure repository/bank for other research studies in the future. If you do not agree to allow this use of your data and/or specimen for future studies approved by the required committees, such as the Institutional Review Board, you will not be able to participate in this study. |
| <b>DISCLOSURE:</b> The VA research team may need to disclose the information listed above to other people or institutions that are not part of VA. VA/VHA complies with the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA), Privacy Act of 1974 and all other applicable federal laws and regulations that protect your privacy. The VHA Notice of Privacy Practices (a separate document) provides more information on how we protect your information. If you do not have a copy of the Notice, the research team will provide one to you. |
| Giving your permission by signing this authorization allows us to disclose your information to other institutions or persons as noted below. Once your information has been disclosed outside VA/VHA, it may no longer be protected by federal laws and regulations and might be re-disclosed by the persons or institutions receiving the information. |
| □ Non-VA Institutional Review Board (IRB) at who will monitor the study |
| Study Sponsor/Funding Source: Veterans Administration VA or non-VA person or entity who takes responsibility for; initiates, or funds this study |
| ☐ Academic Affiliate (institution/name/employee/department): A relationship with VA in the performance of this study |
| Compliance and Safety Monitors: Advises the Sponsor or PI regarding the continuing safety of this study |
| ☐ Other Federal agencies required to monitor or oversee research (such as FDA, OHRP, GAO): |
| ☐ A Non-Profit Corporation (name and specific purpose): |
| ☐ Other (e.g. name of contractor and specific purpose): |


| Authorization for Use & Release of Individually Idea Veterans Health Administration (V | |
|---|---|
| Subject Name (Last, First, Middle Initial): | Subject SSN (last 4 only): Date of Birth: |
| <b>Note:</b> Offices within VA/VHA that are responsible for oversight of VA Oversight (ORO), the Office of Research and Development (ORD), the Office of General Counsel, the VA IRB and Research and Development information in the performance of their VA/VHA job duties. | e VA Office of Inspector General, the VA |
| Access to your Individually Identifiable Health Information create While this study is being conducted, you | ed or obtained in the course of this research |
| ☐ will have access to your research related health records | |
| ⊠ will not have access to your research related health records | |
| This will not affect your VA healthcare including your doctor's ability to and will not affect your right to have access to the research records a | · |
| <b>REVOCATION:</b> If you sign this authorization you may change your m any time. You must do this in writing and must send your written requ the following address: | • |
| Mark Ilgen, PhD<br>VA Ann Arbor Healthcare System<br>2215 Fuller Rd.<br>Ann Arbor, MI 48105 | |
| If you revoke (take back) your permission, you will no longer be able to which you are entitled will NOT be affected. If you revoke (take back) continue to use or disclose the information that it has already collected permission which the research team has relied upon for the research, it is received by the study's Principal Investigator. | your permission, the research team may d before you revoked (took back) your |
| <b>EXPIRATION:</b> Unless you revoke (take back) your permission, your a your information will: | authorization to allow us to use and/or disclose |
| ⊠ Expire at the end of this research study | |
| ☐ Data use and collection will expire at the end of this research study. Any repository to be used for future research will not expire. | study information that has been placed into a |
| ☐ Expire on the following date or event: | |
| ☐ Not expire | |


| Signature of Legal Representative (if applicable) To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
|---|
| Research Subject Signature. This permission (authorization) has been explained to me and I have been given the opportunity to ask questions. If I believe that my privacy rights have been compromised, I may contact the VHA facility Privacy Officer to file a verbal or written complaint. I give my authorization (permission) for the use and disclosure of my individually identifiable health information as described in this form. I will be given a signed copy of this form for my records. Signature of Research Subject Date To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
| opportunity to ask questions. If I believe that my privacy rights have been compromised, I may contact the VHA facility Privacy Officer to file a verbal or written complaint. I give my authorization (permission) for the use and disclosure of my individually identifiable health information as described in this form. I will be given a signed copy of this form for my records. Signature of Research Subject Date To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
| Signature of Research Subject Signature of Legal Representative (if applicable) To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
| Signature of Legal Representative (if applicable) To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
| To Sign for Research Subject (Attach authority to sign: Health Care Power of Attorney, Legal Guardian appointment or Next of Kin if authorized by State Law) |
| Name of Legal Representative (please print) |

## VA INFORMED CONSENT PROCESS CHECKLIST

\*Complete this checklist for each consent obtained and file with the original informed consent document\*

| RESEARCH STUDY IDENTIFICATION (Required information) |
|---|
| STUDY TITLE: Link Up: Facilitating use of the Veterans Crisis Line in High-Risk Patients |
| PI:E. Brooke Pope, PhD |
| NAME OF STUDY TEAM MEMBER OBTAINING CONSENT: |
| ROLE OF STUDY TEAM MEMBER OBTAINING CONSENT: |

ORIGINAL FORM VERSION: 4/15/09. REVISIONS: 9/17/09, 10/30/09, 11/30/09, 12/07/11, 2/27/12, 10/7/13

| RESI | EARCH SUBJECT IDENTIFICAT | ION: (Requir | ed information) | | |
|---|---|---|---|---|---|
| | | | 1 1 1 | 1 1 | |
| Last Name | First Name | Mid. Init. | Last-4 SSN | Todays Date (mm/dd/yy) | _ |

| A. | Date ALL required SIGNATURES (Subject, Witness (If required by IRB) and Person Obtaining |
|---|---|
| | Consent), their PRINTED NAMES and the DATES they signed the informed consent document |
| | (ICD) have been Checked and Verified Accurate and appear in the proper location |
| B. | |
| | DATE AND TIME (ICD) WAS REVIEWED AND DEEMED COMPLETE AND VALID |
| | **Must be prior to date/time of Subject's First Study Activity** |
| C. | |
| | DATE AND TIME OF THE SUBJECT'S FIRST STUDY ACTIVITY OR INVOLVEMENT |
| | Verify and Initial each requirement below. |
| 1. | Informed consent and HIPAA Authorization, if required by VA-IRB was obtained from this |
| | subject prior to study participation. |
| 2. | A VA Scope of Practice Form has been signed by the PI and approved by the VA IRB which |
| | designates me as an authorized agent of the PI and qualified to obtain consent for this study. |
| 3. | This prospective subject was given adequate time necessary to carefully and fully read the |
| | Informed consent document (ICD) and all questions were answered to his/her satisfaction. |
| 4. | All aspects of this subject's study involvement, including the purpose of the study, known and |
| | potential risks, possible benefits and alternatives to study participation were explained and |
| | discussed prior to subject signing the ICD. |
| 5. | If required, a scanned image of the Research Enrollment Note, Consent Form and/or HIPAA |
| | Authorization will be entered into the subject's electronic medical record (CPRS). |
| 6. | Subject has been consented using the most recently approved, VA date-stamped version of |
| | the consent form (VA Form 10-1086) and HIPAA Authorization Form (VA Form 10-0493). |
| 7. | A copy of the completed and signed, original informed consent document has been issued to |
| | this subject and the subject was instructed to retain that copy for reference and to ask any and |
| | all questions that might arise throughout their study involvement. |
| 8. | The subject has been shown where in the ICD to locate study team phone number(s) and the |
| | phone number of the VAAAHS IRB Coordinator. The subject has been reminded to call with any |
| | questions or concerns. Cathy Kaczmarek @ 734.845.3439 |
| 9. | The subject has been informed that participation is entirely voluntary and that they may |
| | withdraw their participation at any time and for any reason. |
| 10. | Original ICDs and all copies are printed and issued as single-sided documents and that the |
| | original signed ICD must be kept in the investigator's project files on VA property. |
| 11. | Upon completion of the Informed Consent Process, this subject's name was added to the |
| | Master List of All Subjects. [Per revised VHA Handbook 1200.05 (11/12/14) a MLS is no |
| | longer required, but a list of all enrolled participants is considered good research practice.] |
| 12. | I know I can contact the VAAAHS IRB Coordinator at 734.845.3439 or the Research |
| | Compliance Officer at 734.845.3766 if I have questions or concerns regarding the consent of |
| | this or any individual considering study participation. |
| | Titles of any individual considering study participation. |



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: E. Brooke Pope, PhD VAMC: Battle Creek VA Healthcare System


### PURPOSE OF RESEARCH STUDY:

The purpose of the study is to learn about Veterans who use the Veterans Crisis Line during a suicidal crisis and those who don't. We would also like to learn whether or not Veterans who have experienced a suicidal crisis could benefit from participating in a discussion about their thoughts and perceptions of the Veterans Crisis Line. You have been invited to participate in this research study because you are a patient in this VA psychiatry inpatient unit and were identified as having experienced a suicidal crisis (i.e. recent suicide attempt, significant suicidal thoughts). This is a joint study between the Battle Creek and Ann Arbor VA facilities.

#### DESCRIPTION:

This is a two part study. Part 1 involves completing a survey only. Based on some of your answers you may be eligible to participate in Part 2. Below is more detail about Part 1 and Part 2:

Part 1: We plan to enroll up to approximately 1042 patients for Part 1 – Screening of this study. If you decide to participate, we will ask you to complete a screening survey, which will take approximately 15-30 minutes. The survey asks questions about topics such as your thoughts and behaviors related to suicide, overall mental health and physical functioning, and your utilization of treatment services, such as the Veterans Crisis Line. Depending on your answers to the screening survey, you may be eligible to participate in the full study (Part 2. If you are found not eligible for participation in the full study, then your participation will be complete at the end of Part 1 and you will have no further contact with our research staff.

Part 2: We plan to enroll approximately 500 patients for Part 2 of this study. If you are eligible and decide to participate in the full study, you will be asked to complete the following:

Baseline Assessment: The baseline assessment will take approximately 45-60 minutes to complete. We will ask questions about topics such as suicide, drug and alcohol use, treatment and service utilization, and perception of those services. You will complete part of the assessment yourself by answering questions on a paper survey and the other part will include interview questions asked by research staff.

*Intervention session:* After completing the baseline assessment you will be randomly placed into one of two groups (assigned by chance in a process similar to "flipping a coin"):

<u>Group 1</u>: If you are in Group 1, you will be asked to participate in a 30-45 minute one-on-one intervention session with a member of our study team to discuss the Veterans Crisis hotline. These sessions will be audio recorded and reviewed by research staff for training purposes and to ensure that the research team is following protocol (making sure that all research team members conduct the sessions in the same way).

<u>Group 2</u>: If you are in Group 2, you will be asked to participate in a brief discussion with a member of our study team, and you will receive informational materials about the Veterans Crisis Line.

Afterwards both groups will be asked to answer some additional questions, which will take approximately 5-10 minutes.

| RESEARCH SUBJECT IDENTIFICATION: (Required information) | | | | | _ |
|---|---|---|---|---|---|
| | | | 1 1 1 | 1 1 | |
| Last Name | First Name | Mid. Init. | Last-4 SSN | Todays Date (mm/dd/yy) | _ |
| VA Form 10-1086 | Page 1 | of 5 | | | |



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: E. Brooke Pope, PhD VAMC: Battle Creek VA Healthcare System


Follow-Up Assessments: Study staff still will contact you to schedule your follow up assessments at about 3, 6, and 12-months after study enrollment. These follow-up sessions will usually take approximately 45-60 minutes. The assessments will ask similar questions as the baseline assessment

Your total participation in Part 2 of the study (i.e. baseline survey, intervention, and 3 follow-up surveys) is expected to occur over a period of approximately 12 months. After you complete the study, we may contact you for an additional interview to ask about your study experience. If you choose to participate in the interview, you will sign a separate consent form for that part.

#### RISKS:

You may experience some discomfort when answering questions, such as questions regarding your experiences with suicide and suicidal thoughts. This type of discomfort is expected to be temporary. You may choose not to answer any questions that make you uncomfortable or that you do not wish to answer.

Another risk is potential loss of confidentiality of some of your personal information. We may be required to break confidentiality if we believe that there is a risk of harm to yourself or someone else (for example, you may harm yourself, someone else, or someone is harming you, or in cases of child or elder abuse). This means that we may be required to inform your regular care providers or authorities to protect you or others. The information we disclose will be relevant to your care and may have been information we obtained during the research, such as your thoughts to harm yourself, your name, and contact information,

As with any research study, there may be other risks that are unforeseeable at this time.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate of Confidentiality does not prevent the researchers from disclosing voluntarily, without your consent, information that would identify you as a participant in the research project under the following circumstances: if you disclose intent to hurt yourself, others, or if you are being hurt.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to get research information, then the researchers may not use the Certificate to withhold that information.



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: E. Brooke Pope, PhD VAMC: Battle Creek VA Healthcare System


Being in more than one research study at the same time, or even at different times, may increase the risks to you. It may also affect the results of the studies. You should not take part in more than one study without approval from the researchers involved in each study.

## **BENEFITS:**

Your participation may help us discover how to improve services for veterans in the future. If you participate in Part 2, you may find that participating in this study helps you to learn about options you may have for obtaining help when in a suicidal crisis. However, we cannot and do not guarantee or promise that you will benefit by participating in this study.

### ALTERNATE COURSES OF ACTION:

You do not have to participate in this study. You may withdraw from the study at any time without penalty. By doing so, you will not lose any benefits that you may be entitled to. If you choose not to participate in this study, your decision will not affect your eligibility to receive standard health care at the Battle Creek VAMC.

## STATEMENT OF RESEARCH RESULTS:

Research data collected as part of this study will be stored according to the privacy and security guidelines established by the VHA. Only authorized research staff will have access to your research data and research files. These authorized research staff may have access to viewing your paper forms and medical records. If you participate in Part 2, authorized research staff may also access your medical records to obtain your contact information to schedule and conduct follow-up appointments. Your name and other identifying information (consent form) will be stored separately from research data (e.g. survey and interview answers). Unique ID numbers will be substituted for names to protect your identity in the data file. Data on paper will be stored in locked filing cabinets at Ann Arbor VA research offices. All electronic study data will be kept in restricted access files and stored on the VA network server. Paper files may be stored on the secure network drive as a PDF. Because this is a joint study between the Battle Creek VAMC and Ann Arbor VAMC, electronic data may be shared/transmitted through the use of VAMC secure servers at either site.

If you participate in Part 2, the audiotapes of the sessions will be converted into computer files and stored on secure servers. Audio-records will be used to evaluate the research staff who are leading the sessions. Audio computer files will be confidential and access will be limited to authorized research staff.

Researchers from the Battle Creek Health Care System and the Ann Arbor VA Health Care System will analyze the data collected from this study. If the results of this study are reported in medical journals or at meetings, you will not be identified by name, by recognizable photograph, or by any other means without your specific consent. No information by which you can be identified will be released or published unless required by law. We will let you know of any important discoveries made during this study which may affect you, your condition, or your willingness to participate in this study.

#### SPECIAL CIRCUMSTANCES:

There will not be any costs to you for any additional care that your receive as a participant in this research study. The investigators of this study may have to end your participation in this study for reasons such as if it is in your best interest; you do not follow the study plan (e.g., do not complete the survey); the investigator



**Title of Study:** Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients

Principal Investigator: E. Brooke Pope, PhD VAMC: Battle Creek VA Healthcare System


decides that continuation could be harmful to you; the study is canceled; other administrative reasons; or other unanticipated circumstances. If you are withdrawn from the study, it will not affect the treatment you receive from your providers at the Battle Creek VAMC.

## **COMPENSATION:**

For participating in Part 1, you will receive a \$10 gift card after completing the screening survey.

If you are eligible after screening, and you choose to participate in Part 2, you will receive a \$25 gift card for completion of the baseline assessment and a \$30 gift card for each 3, 6, and 12 month follow-up assessment completed. Therefore, your maximum compensation for this part of the study could be \$115.



| Title of Study: | Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients | | |
|---|---|---|---|
| Principal Investi | pal Investigator: E. Brooke Pope, PhD VAMC: Battle Creek VA Healthcare System | | |
| RESEARCH SUB | JECT'S | | |
| treatment have been | n explain | has explained this research possible benefits of the study have been des ed. Some veterans are required to pay co-pa syment requirements will continue to apply for | syments for medical care and services |
| no penalty or loss of<br>time without penalty<br>accordance with ap-<br>injured by participat<br>been made for addit<br>medical care and se-<br>care and services p | f rights to<br>or loss of<br>plicable foi<br>ion in this<br>tional cor<br>ervices provided b | entirely voluntary. You may refuse to participe which individuals are entitled. Participants of VA or other benefits. VA will provide treatrederal regulations. The VA will provide neces study. You will be treated for the injury at many mensation. You may be among the veterans to ovided by VA. These co-payment requirements by VA that are not part of this study. You have gents from liability for negligence by signing the study. | may withdraw from this study at any ment for research related injury in ssary medical treatment should you be to cost to you, but no provisions have a required to pay co-payments for the medical enot waived any legal rights or |
| research study, you<br>5600 extension 316<br>after hours at 734-9<br>contacted at 269-96 | can conf<br>34 during<br>36-6266<br>6-5600 e<br>(8255), a | oblems, an injury, or if you have questions, cated member(s) of the research study team: East member(s) of the research study team: East the day. Mark Ilgen can be called at 734-84 (then dial page ID: 15912) or the Battle Creextension 33857 after hours. At any time, you and press "1" to connect to a free, 24-hour VA stration. | Brooke Pope can be called at 269-966-<br>5-3646 during the day and or paged<br>k VA psychiatrist on call can be<br>may call the Veterans Crisis Hotline |
| research subject an study staff are not a | d to verify<br>vailable o | nan Studies coordinator at 734-845-3440 to a this study is reviewed and approved by the or to discuss your questions or concerns with rch at the Battle Creek VA and Ann Arbor V | VA. You may also call when research someone other than study staff. You |
| I have been informe<br>I will receive a signe | | my rights as a research subject, and I volunta<br>f this consent form. | arily consent to participate in this study. |
| Х | | X | x |
| X<br>Signature of Subjec | t | X<br>(Print Name) | Todays Date (mm/dd/yy) |
| • | | , | |
| Х | | X | x |
| XSignature of person<br>(Study personnel must be | | | X<br>Todays Date (mm/dd/yy) |
| IF MORE THAN ONE PAGE IS USED, EACH PAGE (VAF 10-1086) MUST BE CONSECUTIVELY NUMBERED. | | | |
| VA Form 10-1086<br>[VALID ONLY WITH CURF | | Page 5 of 5 | |

| Department of Veterans Affairs Authorization for Use and Release of Individually Identifiable Health Information Collected for VHA Research | | |
|---|---|---|
| Subject Name (Last, First, Middle Initial): | Subject SSN (last 4 only): | Date of Birth: |
| VA Facility (Name and Address): Battle Creek VA Medical Center 5500 Armstrong Road Battle Creek, MI 49037-7314 | | |
| VA Principal Investigator (PI): | PI Contact Information: | |
| E. Brooke Pope, Ph.D. | Elizabeth.Pope2@va.gov; 269-966-5600 x31634 | |
| Study Title: | 1 | |
| Link Up: Facilitating Use of the Veterans Crisis Line in High-Risk Patients | | |
| Purpose of Study: The purpose of the study is to learn about Veterans who use the Veterans Crisis Li also like to learn whether or not Veterans who have experienced a suicidal crisis of member of our study team about their thoughts and perceptions of the Veterans Crisearch study because you are a patient in this VA psychiatry inpatient unit and we recent suicide attempt, significant suicidal thoughts). Based on your responses proinvited to participate in further research activities, including further surveys, interviolet (Part 2). This is a joint study between the Battle Creek and Ann Arbor VA facilities. | ould benefit from participating in a drisis Line. You have been invited to pare identified as having experienced vided during the screening survey (Paviews and a discussion with a member | iscussion with a participate in this a suicidal crisis (i.e. art 1), you may be |
| USE OF YOUR INDIVIDUALLY IDENTIFIABLE HEALTH INFORM | MATION (IIHI): | |
| Your individually identifiable health information is information about information that would identify you such as your name, date of birth to allow the VA Principal Investigator (PI) and/or the VA research to present health information in addition to new health information the investigators of this study are committed to protecting your privacy your health care. | n, or other individual identifiers.<br>eam members to access and u<br>ov may collect for the study nan | . VHA is asking you<br>ise your past or<br>ned above. The |
| Signing this authorization is completely voluntary. However, your are participate in this study. Your treatment, payment, enrollment, or el whether or not you sign this authorization. | igibility for VA benefits will not | be affected, |
| Your individually identifiable health information used for this VA stu | dy includes the information ma | arked below: |
| $oxed{\boxtimes}$ Information from your VA Health Records such as diagnoses, findings | progress notes, medications, | lab or radiology |
| Specific information concerning: | | |
| $oxed{oxed}$ alcohol abuse $oxed{oxed}$ drug abuse $oxed{oxed}$ sickle cell | I anemia | |
| ☑ Demographic Information such as name, age, race | | |
| ☐ Billing or Financial Records | | |
| <ul> <li>☑ Questionnaire, Survey, and/or Subject Diary</li> <li>☑ Other as described: We will only access information concerning alcohol or</li> </ul> | or drug abuse for participants in Part | 2. |

**Version Date:** 06/0<u>9</u>/2016


| Veterans Health Administration (VHA) Research Subject Name (Last, First, Middle Initial): Subject SSN (last 4 only): Date of Birth: |
|---|
| Subject Name (Last, 1 list, whome milial). |
| USE OF YOUR DATA OR SPECIMENS FOR OTHER RESEARCH: (Instruction: When banking or further analysis is an optional research activity, complete page 5 and leave this section blank. If banking is a required research activity to store "Data" and/or "Specimen" for future use or if "Not Applicable" is selected, remove page 5 in its entirety.) |
| An important part of this research is to save your |
| □ Data |
| ☐ Specimen |
| in a secure repository/bank for other research studies in the future. If you do not agree to allow this use of your data and/or specimen for future studies approved by the required committees, such as the Institutional Review Board, you will not be able to participate in this study. |
| <b>DISCLOSURE:</b> The VA research team may need to disclose the information listed above to other people or institutions that are not part of VA. VA/VHA complies with the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA), Privacy Act of 1974 and all other applicable federal laws and regulations that protect your privacy. The VHA Notice of Privacy Practices (a separate document) provides more information on how we protect your information. If you do not have a copy of the Notice, the research team will provide one to you. |
| Giving your permission by signing this authorization allows us to disclose your information to other institutions or persons as noted below. Once your information has been disclosed outside VA/VHA, it may no longer be protected by federal laws and regulations and might be re-disclosed by the persons or institutions receiving the information. |
| □ Non-VA Institutional Review Board (IRB) at who will monitor the study |
| Study Sponsor/Funding Source: Veterans Administration VA or non-VA person or entity who takes responsibility for; initiates, or funds this study |
| ☐ Academic Affiliate (institution/name/employee/department): A relationship with VA in the performance of this study |
| Compliance and Safety Monitors: Advises the Sponsor or PI regarding the continuing safety of this study |
| ☐ Other Federal agencies required to monitor or oversee research (such as FDA, OHRP, GAO): |
| ☐ A Non-Profit Corporation (name and specific purpose): |
| ☐ Other (e.g. name of contractor and specific purpose): |


| Authorization for Use & Release of Individually Idea Veterans Health Administration (V | |
|---|---|
| Subject Name (Last, First, Middle Initial): | Subject SSN (last 4 only): Date of Birth: |
| <b>Note:</b> Offices within VA/VHA that are responsible for oversight of VA Oversight (ORO), the Office of Research and Development (ORD), the Office of General Counsel, the VA IRB and Research and Development information in the performance of their VA/VHA job duties. | ne VA Office of Inspector General, the VA |
| Access to your Individually Identifiable Health Information create While this study is being conducted, you | ed or obtained in the course of this researc |
| ☐ will have access to your research related health records | |
| ⊠ will not have access to your research related health records | |
| This will not affect your VA healthcare including your doctor's ability to and will not affect your right to have access to the research records at | |
| <b>REVOCATION:</b> If you sign this authorization you may change your many time. You must do this in writing and must send your written require the following address: | • • |
| E. Brooke Pope, PhD Battle Creek VA Medical Center 5500 Armstrong Road Battle Creek, MI 49037-7314 | |
| If you revoke (take back) your permission, you will no longer be able to which you are entitled will NOT be affected. If you revoke (take back) continue to use or disclose the information that it has already collected permission which the research team has relied upon for the research, it is received by the study's Principal Investigator. | your permission, the research team may d before you revoked (took back) your |
| <b>EXPIRATION:</b> Unless you revoke (take back) your permission, your a your information will: | authorization to allow us to use and/or disclose |
| ⊠ Expire at the end of this research study | |
| ☐ Data use and collection will expire at the end of this research study. Any repository to be used for future research will not expire. | study information that has been placed into a |
| ☐ Expire on the following date or event: | |
| ☐ Not expire | |


| Authorization for Use & Release of Individually Identifiable Health Information for<br>Veterans Health Administration (VHA) Research | | |
|---|---|---|
| Subject Name (Last, First, Middle Initial): | Subject SSN (last 4 only): | Date of Birth: |
| TO BE FILLED OUT BY THE S | SUBJECT | |
| Research Subject Signature. This permission (authorization) has be opportunity to ask questions. If I believe that my privacy rights have be facility Privacy Officer to file a verbal or written complaint. | | |
| I give my authorization (permission) for the use and disclosure of my described in this form. I will be given a signed copy of this form for my | | h information as |
| Signature of Research Subject | Date | |
| Signature of Legal Representative (if applicable) | Date | _ |
| To Sign for Research Subject (Attach authority to sign: Health Care F or Next of Kin if authorized by State Law) | Power of Attorney, Legal Gua | ardian appointment, |
| Name of Legal Representative (please print) | | |